CLINICAL TRIAL: NCT01260779
Title: Open Label Expanded Access for Investigational Use of PV-10 in Patients Who Are Not Eligible for an Existing PV-10 Clinical Trial, for Whom There is no Alternative Therapy, and Whom May Benefit From PV-10 Administration
Brief Title: Expanded Access Protocol for PV-10 for Cutaneous or Subcutaneous Tumors
Status: No longer available | Type: Expanded Access
Sponsor: Provectus Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Provectus Pharmaceuticals (Industry)
Other Study IDs: PV-10-EA-02
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Cutaneous or Subcutaneous Tumors Where There is no Comparable or Satisfactory; Approved Alternative Therapy
MeSH Terms: interventions — Rose Bengal

INTERVENTIONS:
Drug: PV-10 (10% rose bengal disodium) — Intralesional injection for chemoablation of cutaneous or subcutaneous lesions

SUMMARY:
This compassionate use protocol provides expanded access for investigational use of PV-10 in cancer patients who are not eligible for an existing PV-10 clinical trial, for whom there is no comparable or satisfactory approved alternative therapy and whom, in the opinion of the investigator, may benefit from PV-10 administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, male or female.
2. Histologically or cytologically confirmed cancer where there is no comparable or satisfactory approved alternative therapy specific to cutaneous or subcutaneous tumors.
3. Performance Status: ECOG 0-2.
4. Life Expectancy: At least 6 months.
5. Blood Chemistry:

   * Creatinine ≤ 3 times the upper limit of normal (ULN).
   * Total bilirubin ≤ 3 times the upper limit of normal (ULN).
   * AST/ALT/ALP ≤ 5 times the upper limit of normal (ULN).
6. Thyroid Function

   * Total T3 or free T3 (serum triiodothyronine), total T4 or free T4 (serum thyroxine) and THS (serum thyrotropin) ≤ grade 2 abnormality.
7. Renal Function

   * Subjects must have adequate renal function in the opinion of the Investigator with no clinically significant renal impairment or uncontrolled renal disease.

Exclusion Criteria:

1. Cancer patients who are eligible for an existing PV-10 clinical trial.
2. Certain photosensitizing agents within 5 half-lives prior to PV-10 administration.
3. Concurrent or Intercurrent Illness:

   * Subjects with uncontrolled diabetes or extremity complications due to diabetes.
   * Subjects with severe peripheral vascular disease.
   * Subjects with significant concurrent or intercurrent illness, psychiatric disorders, or alcohol or chemical dependence that would, in the opinion of the Investigator, compromise their safety or compliance or interfere with interpretation of study results.
   * Subjects with uncontrolled thyroid disease, goiter, partial thyroidectomy, radioiodine- or surgically-treated Graves' hyperthyroidism or cystic fibrosis.
   * Subjects with clinically significant acute or unstable cardiovascular, (stroke), renal, gastrointestinal, pulmonary, immunological (with the exception of the presence of hepatitis B virus (HBV), viral hepatitis, or cirrhosis), endocrine, or central nervous system disorders.
4. Pregnancy:

   * Female subjects who are pregnant or lactating.
   * Female subjects who have positive serum ßHCG pregnancy test taken within 7 days of PV-10 administration.
   * Fertile subjects who are not using effective contraception.
5. Investigational Agents:

   * Subjects who have received investigational agents within 4 weeks (or 5 half-lives) of study administration.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - St Luke's University Health Network, Bethlehem, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Melanoma Institute Australia, Sydney (North Sydney and Camperdown), New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital Cancer Centre, Adelaide, South Australia